CLINICAL TRIAL: NCT05529381
Title: Anxiety and Depressive Symptoms of Pregnant Women Diagnosed to Have Placenta Previa / Accreta
Brief Title: Anxiety and Depressive Symptoms in Placenta Previa / Accreta
Status: Completed | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, AM Abdelbary, principle investigator, Assiut University
Other Study IDs: ADSPPP
Record Dates: First submitted 2022-09-02; First posted 2022-09-07 (Actual); Last update posted 2024-11-08 (Actual); Status verified 2024-02

CONDITIONS: Anxiety Depression; Placenta Previa
MeSH Terms: conditions — Placenta Previa

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
placenta previa is an obstetric complication which is associated with depression and anxiety.

As little is known about the emotional reaction to the diagnosis of placenta previa/accrete, a study is badly needed to estimate the magnitude of this problem and its effects on the mother

DETAILED DESCRIPTION:
Placenta previa is an obstetric complication with a prevalence of 5.2 per 1000 pregnancies. placenta previa is associated with maternal morbidity and mortality. The delivery carries a risk of bleeding, emergency hysterectomy, organ damage and even death. During admission, counselling is done for the possible need for delivery at any time and the need for life saving hysterectomy. hysterectomy is a tough and difficult choice for patients, and the subsequent emotional process is often associated with depression, severe and prolonged feelings of sadness, diminished interest in activities and in sexual intercourse. Similarly, severe adverse psychological outcomes, including post-traumatic stress disorders, have been reported as a result of traumatic birth events. Antenatal depression and anxiety occur in approximately 13% and up to 21.7% of women, respectively. Rates of antenatal depression among women hospitalized for obstetrical risk can be as high as 19%.

Research about the responses to a diagnosis of placenta previa is scarce. A study found increased anxiety score in women diagnosed with Placenta accreta spectrum. Other studies focussed on the post-trauma stress associated with hysterectomy versus uterine conservation.

As little is known about the emotional reaction to the diagnosis of placenta previa/accrete, a study is badly needed to estimate the magnitude of this problem and its effects on the mother.

ELIGIBILITY:
Inclusion Criteria:

* patient diagnosed to have placenta previa or accrete
* plan to deliver baby in Assiut women health hospital
* willing and able to participate

Exclusion Criteria:

* pre-existing psychological disorders
* severe medical complications
* severe obstetric complications
* fetal abnormality

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes
Study Population: pregnant women diagnosed to have placenta previa / accreta in Inpatient ward Assuit women health hospital
Sampling Method: Non-Probability Sample
Enrollment: 73 (Actual)
Dates: Start 2022-11-26 (Actual); Primary Completion 2024-06-06 (Actual); Study Completion 2024-11-06 (Actual)

PRIMARY OUTCOMES:
Assess stress, anxiety and depression symptoms in inpatients diagnosed to have placenta previa /accreta | 5 minutes
  Depression Anxiety Stress Scale-21

SECONDARY OUTCOMES:
Effects of depressive and anxiety symptoms on women functioning and quality of life | 10 minutes
  SF-12 questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut University, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Byatt N, Hicks-Courant K, Davidson A, Levesque R, Mick E, Allison J, Moore Simas TA. Depression and anxiety among high-risk obstetric inpatients. Gen Hosp Psychiatry. 2014 Nov-Dec;36(6):644-9. doi: 10.1016/j.genhosppsych.2014.07.011. Epub 2014 Jul 27. PMID 25149040
- [Background] Crocetto F, Barone B, Bonito E, Maggi M, Caputo VF, di Girolamo A, Trama F, di Spiezio Sardo A, Zizolfi B. Psychological impact of abnormally invasive placenta: an underestimated and hidden morbidity. J Basic Clin Physiol Pharmacol. 2022 Apr 8;33(5):649-653. doi: 10.1515/jbcpp-2021-0384. eCollection 2022 Sep 1. PMID 35388654
- [Background] Jenabi E, Salimi Z, Bashirian S, Khazaei S, Ayubi E. The risk factors associated with placenta previa: An umbrella review. Placenta. 2022 Jan;117:21-27. doi: 10.1016/j.placenta.2021.10.009. Epub 2021 Oct 20. PMID 34768164
- [Background] Lovibond PF, Lovibond SH. The structure of negative emotional states: comparison of the Depression Anxiety Stress Scales (DASS) with the Beck Depression and Anxiety Inventories. Behav Res Ther. 1995 Mar;33(3):335-43. doi: 10.1016/0005-7967(94)00075-u. PMID 7726811
- [Background] Park HS, Cho HS. Management of massive hemorrhage in pregnant women with placenta previa. Anesth Pain Med (Seoul). 2020 Oct 30;15(4):409-416. doi: 10.17085/apm.20076. PMID 33329843
- [Background] Tol ID, Yousif M, Collins SL. Post traumatic stress disorder (PTSD): The psychological sequelae of abnormally invasive placenta (AIP). Placenta. 2019 Jun;81:42-45. doi: 10.1016/j.placenta.2019.04.004. Epub 2019 Apr 16. PMID 31138430
- See also: Related Info — http://www.physio-pedia.com/12-Item_Short_Form_Survey_(SF-12)